CLINICAL TRIAL: NCT02358954
Title: Modulation of Pain Responses by Vestibular Stimulation. A Contact Heat Evoked Potential Study.
Brief Title: Vestibular Pain Interactions
Acronym: VPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Lucian Macrea, Lucian M Macrea, University of Zurich
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VPI01
Record Dates: First submitted 2015-01-22; First posted 2015-02-09 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: quantitative sensory testing; contact heat evoked potentials; vection stimulation; 3D-turntable; Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vestibular Pain interactions (Experimental)
  Interventions: Procedure: Quantitative sensory testing; Procedure: CHEPS; Procedure: 3D Turntable; Procedure: Vection stimulation

INTERVENTIONS:
Procedure: Quantitative sensory testing — Measurement of warm and cold detection and pain thresholds
  Other Names: QST
Procedure: CHEPS — Measurement of amplitude and latency of cortically evoked potentials
  Other Names: Contact heat evoked potentials
Procedure: 3D Turntable
Procedure: Vection stimulation

SUMMARY:
The goal is to establish the practical usefulness of vestibular stimulation for modulating pain perception and to describe the possible mechanisms that could underlie neural vestibular-somatosensory interactions.

ELIGIBILITY:
Inclusion Criteria:

* Weight: 50 - 100 kg
* Height: 155 - 185 cm
* Male subjects 18 years to 60 years of age
* Sufficient command of German language
* Written informed consent by the participant after information about the project
* Without any known history of neurological disease (especially motor, somatosensory disorders, peripheral neuropathies).
* Right-handedness

Exclusion Criteria:

1. Intellectually or mental impaired subjects
2. Drug abuse
3. Chronic alcohol consumption
4. No use of marihuana 24h before measurements.
5. No history of vestibular or auditory disorders.
6. Diabetes mellitus
7. Participants of other studies during study period and 30 days prior to study begin
8. Any regular concomitant medication
9. Abnormal QST parameters at the baseline measurement.
10. Absent CHEPs-Potentials at the baseline measurement.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pain thresholds | After study inclusion, Day1
  The change in heat or cold pain threshold after physical vestibular stimulation and vection stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Zurich, Zurich, Canton of Zurich, Switzerland